CLINICAL TRIAL: NCT02082145
Title: Electrical Stimulation in Diabetic Peripheral Neuropathy
Acronym: NERVES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13/LO/1844; 13HH1825 (Other: Imperial College London)
Record Dates: First submitted 2014-01-09; First posted 2014-03-10 (Estimated); Results first posted 2019-10-11 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: NMES; Control
Keywords: NMES; diabetic peripheral neuropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Treated according to local protocol for diabetic peripheral neuropathy
- NMES (Experimental): Treated with neuromuscular stimulation of both legs, for 10 weeks
  Interventions: Device: NMES

INTERVENTIONS:
Device: NMES — Application of NMES device bilaterally, once a day, 5 times a week, for 10 weeks
  Arms: NMES

SUMMARY:
To assess the effect of the device on the progression of diabetic peripheral neuropathy

DETAILED DESCRIPTION:
Diabetes is a metabolic disease that affects the body's ability to control blood sugar levels. This affects the tissues of the body, particularly the walls of blood vessels. People with diabetes are more likely to suffer from ischaemic heart disease, stroke, kidney problems, blindness, foot ulcers, and peripheral nerve problems. Diabetes affects approximately 347 million people worldwide, and by 2030 the WHO projects that complications of diabetes will be the 7th leading cause of death.

Peripheral neuropathy is a dysfunction of the nerves most commonly affecting the arms and legs. Diabetes is the leading cause of neuropathy in the Western world, and diabetic neuropathy is estimated to affect between 20-50% of diabetic people. The American Diabetes Association define it as the 'presence of symptoms and signs of peripheral nerve dysfunction in patients with diabetes after exclusion of other causes'. As regards complications of diabetes, peripheral neuropathy has the greatest detrimental effect on quality of life. Diabetic neuropathy is implicated in 50-75% of non-traumatic amputations.

The device to be tested mimics the effect of walking by stimulating the motor nerves of the leg, making the foot twitch- it increases blood flow to the limb and exercises the leg muscles. We have seen previous clinical cases of improvement in peripheral neuropathy with use of the device, and wish to formalise the benefits to patients. It is hypothesised to work either by increasing blood flow to the limb and therefore the nerves themselves, or for electrical current to be having a direct effect on the peripheral nervous system itself. The device is easily fitted, can be self-administered by patients, and is suitable for out-patient therapy.

We wish to evaluate both the short- and longer-term effects of a neuromuscular stimulator on diabetic peripheral neuropathy as a therapeutic intervention.

ELIGIBILITY:
Inclusion criteria

* 18+ years old
* Diabetes as defined by WHO diagnostic criteria on best medical therapy
* Diabetic peripheral polyneuropathy present, confirmed by nerve conduction testing

Exclusion criteria

* Pregnancy
* Pacemaker
* Metal implants in the legs (below knee)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A H Davies, Principal Investigator — Imperial College London
Locations (1):
- Academic Vascular Surgery, Charing Cross Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kluding PM, Pasnoor M, Singh R, Jernigan S, Farmer K, Rucker J, Sharma NK, Wright DE. The effect of exercise on neuropathic symptoms, nerve function, and cutaneous innervation in people with diabetic peripheral neuropathy. J Diabetes Complications. 2012 Sep-Oct;26(5):424-9. doi: 10.1016/j.jdiacomp.2012.05.007. Epub 2012 Jun 18. PMID 22717465
- [Background] Balducci S, Iacobellis G, Parisi L, Di Biase N, Calandriello E, Leonetti F, Fallucca F. Exercise training can modify the natural history of diabetic peripheral neuropathy. J Diabetes Complications. 2006 Jul-Aug;20(4):216-23. doi: 10.1016/j.jdiacomp.2005.07.005. PMID 16798472

RESULTS

PARTICIPANT FLOW:
Groups:
- NMES: Treated with neuromuscular stimulation of both legs for 10 weeks
Period: Overall Study
Arm/Group | Control | NMES
Started | 5 | 9
Completed | 5 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | NMES | Total
Number analyzed (Participants) | 5 | 9 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.6 (1) | 65.8 (1) | 69 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 1 | 8 | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 5 | 9 | 14
Insulin dependance [Number; unit: participants] | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Nerve Conduction Speed (Common Peroneal Nerve)
Time Frame: Baseline, 10 weeks
Measure: Mean (Standard Deviation); unit: m/sec
Groups:
- Control (Week 0): week 0 - Treated according to local protocol for diabetic peripheral neuropathy
- Control (Week 10): week 10 - Treated according to local protocol for diabetic peripheral neuropathy
- NMES (Week 0): week 0 - Treated with neuromuscular stimulation of both legs
- NMES (Week 10): week 10 - Treated with neuromuscular stimulation of both legs
Arm/Group | Control (Week 0) | Control (Week 10) | NMES (Week 0) | NMES (Week 10)
Number analyzed (Participants) | 3 | 3 | 3 | 3
m/sec | 33.93 (29.4) | 44.1 (3.2) | 41.63 (0.5) | 44.13 (2.8)

2. Secondary Outcome: PAID - Quality of Life Questionnaires
Description: PAID (Problem Areas in Diabetes) is a self-administered 20-item scale. Each item is scored from 0 (not a problem) to 4 (serious problem). The sum of all item scores multiplied by 1.25 gives the total PAID score, which ranges from 0 to 100, higher scores reflecting greater emotional distress.
Time Frame: Baseline, 10 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control (Week 0) | Control (Week 10) | NMES (Week 0) | NMES (Week 10)
Number analyzed (Participants) | 5 | 5 | 8 | 3
score on a scale | 26.2 (21.23) | 27.4 (21.93) | 40.29 (17.94) | 5 (4.24)

ADVERSE EVENTS:
Time Frame: 10 weeks
Groups:
- NMES: Treated with neuromuscular st8imulation of both legs
Arm/Group | Control | NMES
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/9
Other Adverse Events (participants affected / at risk) | 0/5 | 0/9

LIMITATIONS AND CAVEATS:
Results are limited by both patient availability for nerve conduction studies, and the return of questionnaires. All patients were followed up, and all adverse results were reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes